CLINICAL TRIAL: NCT00419081
Title: A Phase IIb, Multicenter, Open-Label, Nonrandomized, Repeat-Dose Study of Forodesine Hydrochloride in Patients With Relapsed/Refractory Precursor T-Lymphoblastic Leukemia/Lymphoma Who Have Failed Two or More Prior Treatment Regimens.
Brief Title: Study of Forodesine Hydrochloride in Patients With Relapsed/Refractory Precursor T-Lymphoblastic Leukemia/Lymphoma Who Have Failed Two or More Prior Treatment Regimens
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with Manufacturing
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-Tio-05-202
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Leukemia; Lymphoma
Keywords: leukemia; lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

INTERVENTIONS:
Drug: Forodesine Hydrochloride Sterile Solution, 5 mg/mL
Drug: Forodesine Hydrochloride Capsules (100 mg)

SUMMARY:
The purpose of this study is to determine whether Forodesine Hydrochloride is effective in treating patients with relapsed/refractory precursor T-Lymphoblastic Leukemia/Lymphoma who have failed two or more prior treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an unequivocal histologic diagnosis of precursor T-lymphoblastic leukemia/lymphoma (World Health Organization [WHO] classification).
* Failure to have responded to or relapsed after two or more treatment regimens for their disease, one of which could be HSCT.
* Performance status of 2 by Eastern Cooperative Oncology Group (ECOG) criteria (see Appendix A).
* Eighteen years of age and older.
* Life expectancy of at least three months.
* Adequate liver function (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] ≤3 times upper limit of normal), unless related to the underlying leukemia.
* Negative serum or urine pregnancy test within two to seven days prior to the start of study treatment in females of childbearing potential.
* Females of childbearing potential and males must be willing and able to use an adequate method of contraception to avoid pregnancy for the duration of the study in such a manner that the risk of pregnancy is minimized. Acceptable contraceptives include intra-uterine devices (IUDs), hormonal contraceptives (oral, depot, patch, or injectable), and double-barrier methods such as condoms or diaphragms with spermicidal gel or foam.
* Signed informed consent form (ICF) prior to start of any study-specific procedures.
* Willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act (HIPAA) policy (U.S. patients only).

Exclusion Criteria:

* Patients with known human immunodeficiency virus (HIV) infection or human T lymphotrophic virus 1 (HTLV-1).
* Patients with active hepatitis B or C infection.
* Patients with clinical evidence of active central nervous system (CNS) leukemia.
* Active serious infection not controlled by oral or intravenous antibiotics.
* Patients with a calculated creatinine clearance of <50 mL/min.
* Prior treatment with any investigational antileukemic or chemotherapy agent within seven days prior to study entry or lack of full recovery from side effects due to prior therapy, independent of when that therapy was given.
* Rapidly progressive disease with compromised organ function judged to be life threatening by the Investigator.
* Concurrent treatment with other antileukemia agents (CNS prophylaxis [e.g., intrathecal methotrexate, cytarabine, or hydrocortisone] and corticosteroid use will not be excluded, but must first be approved by the Medical Monitor) (see Sections 9.2.1 and 9.2.2).
* Pregnant and/or lactating female.
* Patients who cannot swallow or who have chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the product.
* Hypersensitive or intolerant to any component of the study drug formulations.
* Patients who have received prior forodesine treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the rate of complete remission for T lymphoblastic leukemia/lymphoma relapsed or refractory patients. The complete remission rate will be evaluated over the three-month Initial Treatment Period.

SECONDARY OUTCOMES:
To determine the rate of CR achieved based on prior HSCT status
Assess safety and tolerability
Assess survival end points
Evaluate the maintenance and duration of response
Evaluate the proportion of patients able to proceed to HSCT
Evaluate the effects of this forodesine regimen on plasma levels of dGuo
Determine the effects of this forodesine regimen on clinical end points
Explore potential predictive biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Auro del Giglio, MD, Principal Investigator — Faculdade de Medicina do ABC; Belinda Pinto Simoes, MD, Principal Investigator — Hospital das Clinicas de Faculdade de Medicina de Ribeirao Preto; Carlos Sergio Chiattone, MD, Principal Investigator — Irmandade da Santa Casa de Misercordia de Sao Paulo; Carmino Antonio de Souza, MD, Principal Investigator — Hospital de Clinicias da UICAMP - Centro de Hematologia e Hemoterapia; David Barqueti Jendiroba, MD, Principal Investigator — Centro Goiano de Oncologia; Ernesto de Meis, MD, Principal Investigator — INCA - Instituto Nacional de Cancer; Fernando Antonio Sellos Ribeiro, MD, Principal Investigator — Instituto Estadual de Hematologia Artur de Siqueira Cavalcanti - HEMORIO; Ines Guterres, MD, Principal Investigator — Hospital Nossa Senhora de Conceicao; Johnny Francisco Cordeiro Camargo, MD, Principal Investigator — Hospital Erasto Gaertner - Liga Paranaense de Combate ao Cancer - CEPEP; Jose Salvador Rodrigues Oliveira, MD, Principal Investigator — Hospital Santa Marcelina; Lucia Mariano da Rocha Silla, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Mair Pedro de Souza, MD, Principal Investigator — Fundacao Hospital Amaral Carvalho; Maria Aparecida Zanichelli, MD, Principal Investigator — Hospital Brigadeiro; Maria Lucia de Martino Lee, MD, Principal Investigator — Instituto de Oncologia Pediatrica - GRAACC Grupo de Apoio as Adolescente e a Crianca com Cancer - UNIFESP; Ricardo Pasquini, MD, Principal Investigator — Hospital de Clinicas da Universidade Federal do Parana; Nicholas Novitzky, MD, Principal Investigator — Division of Haematology; Vernon Louw, MD, Principal Investigator — Free State University; Farhad Ravandi, MD, Principal Investigator — M.D. Anderson Cancer Center; Karen Seiter, MD, Principal Investigator — New York Medical College, Division of Oncology; Francesco Turturro, MD, Principal Investigator — Louisana State University Health Sciences Center; Luis Isola, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Wendy Stock, MD, Principal Investigator — University of Chicago Hospital; Francisco Gonzalez, MD, Principal Investigator — Liberty Hematology and Oncology; James Foran, MD, Principal Investigator — University of Alabama at Birmingham; Ellen Ritchie, MD, Principal Investigator — Weill Medical College of Cornell University; Leonard Heffner, MD, Principal Investigator — The Emory Clinic; Madan Jagasia, MD, Principal Investigator — The Vanderbilt University Medical Center; Katarzyna Jamieson, MD, Principal Investigator — University of Florida; Gary Schiller, MD, Principal Investigator — University of California, Los Angeles; Anjali Advani, MD, Principal Investigator — The Cleveland Clinic; Kellie Sprague, MD, Principal Investigator — Tufts Medical Center; Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Meir Wetzler, MD, Principal Investigator — Roswell Park Cancer Institute; Alexander Gaiger, MD, Principal Investigator — Medical University Hospital; Werner Linkersch, MD, Principal Investigator — Department of Heamtology; David Nachbaur, MD, Principal Investigator — Department of Heamatology; Agnes Buzin, MD, Principal Investigator; Stephane de Botton, MD, Principal Investigator; Jacques Delaunnay, MD, Principal Investigator; Herve Dombret, MD, Principal Investigator — Service Clinique des Maladies du Sang; Francoise Huguet-Rigal, MD, Principal Investigator — Service d'Hematologie; Norbert Ifrah, MD, Principal Investigator; Arnaud Pigneux, MD, Principal Investigator — CHU du Hart Leveque; Bruno Quesnel, MD, Principal Investigator; Houmedaly Reman, MD, Principal Investigator; Xavier Thomas, MD, Principal Investigator — Maladies du Sang; Norbert Vey, MD, Principal Investigator; Francis Witz, MD, Principal Investigator; Genadi Iosava, MD, Principal Investigator — Institute for Heamatology & Transfusiology; Mamia Zodelava, MD, Principal Investigator — Heamatology and Transfusiology Dept; Reinhard Andreesen, MD, Principal Investigator — Universitat Regensburg; Walter Aulitzky, MD, Principal Investigator — Innere Abt. II; Ulrich Duehrsen, MD, Principal Investigator; Gerhard Ehninger, MD, Principal Investigator — Klinikum Carl Gustav Carus der Technischen Universitat; Arnold Ganser, MD, Principal Investigator — ABT Hamatologie und Onkologie; R. Haas, MD, Principal Investigator — Universitatsklinik Dusseldorf; Dieter Hoelzer, MD, Principal Investigator — Leiterin der Studienzentrale; W-D Ludwig, MD, Principal Investigator — Charite Universitatsmedizin Berlin; Deiter Niederwieser, MD, Principal Investigator — Abt. Haematologie / Onkologie; Michael Pfreunschuh, MD, Principal Investigator — Medizinische Klinik I; Mathias Schmid, MD, Principal Investigator — Innere Medizin III, Hamatologie und Onkologie; Norbert Schmitz, MD, Principal Investigator — Hamatologsiche Abteilung; Peter Staib, MD, Principal Investigator — Med. Klinik I / Hamatolgie; Matthias Stelljes, MD, Principal Investigator — Innere Medizin A; Michele Baccarani, MD, Principal Investigator — Istitutp di Ematologia ed Oncologia Medica; Renato Bassan, MD, Principal Investigator — Dipartimento di Oncoloia ed Ematico; Alberto Bosi, MD, Principal Investigator — Aziendo Osperdaliero Universitaria Careggi Oncologia; Felicetto Ferrara, MD, Principal Investigator — Azienda Ospedaliera Antonio Cardarelli; Roberto Foa, MD, Principal Investigator — Cattedra di Ematologie; Eugenio Gallo, MD, Principal Investigator — Divisione di Ematologia; Vincenzo Liso, MD, Principal Investigator — UO Universita degi Studi Policinico Ematologia; Salvatore Mirto, MD, Principal Investigator — Azienda Osperdaliera Vincenzo Cervello Divisione; Enrica Morra, MD, Principal Investigator — Complessa di Ematologia and Dir Departmento; Enrico Pogliani, MD, Principal Investigator — Ematologia; Bob Lowenberg, MD, Principal Investigator — Eramus University Medical Centre; Jerzy Holowiecki, MD, Principal Investigator — Klinika Hematologii I; Wieslaw Jedrzejczak, MD, Principal Investigator — Klinika Hematologii i Onkologii; Kazimierz Kuliczkowski, MD, Principal Investigator — Department of Heamatology; Tadeusz Robak, MD, Principal Investigator — Klinika Hematologii Akademii Meduycznej Wojewodzki; Aleksander Skotnicki, MD, Principal Investigator — Katedra i Klinika Hematologii Collegium Medicum; K. Abdulkadyrov, MD, Principal Investigator — Head of Hematology Clinic; Anatoli Golenkov, MD, Principal Investigator — Head of Clinical Heam and Immunotherapy Dept.; S. Moiseev, MD, Principal Investigator — Faculty Therapy Dept; Valerie Savchenko, MD, Principal Investigator — Dir. Research Institute for BMT and Molecular Hematology; J. Ribera, MD, Principal Investigator — Insitut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol
Locations (5):
- United States (5):
  - University of Chicago Medical Center, Chicago, Illinois
  - Louisana State University Health Sciences Center, Shreveport, Louisiana
  - New York Medical College Division of Oncology, Valhalla, New York
  - Liberty Hematology and Oncology, Columbia, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas